CLINICAL TRIAL: NCT02104895
Title: Randomised Phase 3 Trial Of Accelerated Partial Breast Irradiation Using Intensity Modulated Radiotherapy Versus Whole Breast Irradiation
Brief Title: Accelerated Partial Breast Irradiation Using Intensity Modulated Radiotherapy Versus Whole Breast Irradiation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor; Chief Radiotherapy-Oncology Unit; Florence University, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APBI-IMRT-Florence
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Early breast cancer; Adjuvant breast cancer; Accelerated partial breast irradiation; Intensity modulated radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole breast irradiation (WBI) (Active Comparator): Conventional whole breast irradiation (WBI)
  Interventions: Radiation: Whole breast irradiation (WBI)
- Partial breast irradiation (APBI) (Experimental): Accelerated partial breast irradiation (APBI)
  Interventions: Radiation: Accelerated partial breast irradiation (APBI)

INTERVENTIONS:
Radiation: Accelerated partial breast irradiation (APBI) — Accelerated partial breast irradiation (APBI) using intensity modulated radiotherapy (IMRT)
  Arms: Partial breast irradiation (APBI)
Radiation: Whole breast irradiation (WBI) — Conventional whole breast irradiation (WBI)
  Arms: Whole breast irradiation (WBI)

SUMMARY:
The aim of this Phase 3 randomised trial is to compare the efficacy and safety of whole breast radiotherapy to accelerated partial breast irradiation using intensity-modulated radiotherapy technique in selected early breast cancer patients after breast conserving surgery.

DETAILED DESCRIPTION:
The surgeons were requested to place clips at the borders of the surgical bed, using a minimum of four clips. The presence of surgical clips was a selection criterion to avoid geographic misses. Computed tomography (CT) scanning was performed using 0.3-cm thick-slices and a slice spacing of 0.3 cm.

In patients assigned to APBI arm, the clinical target volume (CTV) was drawn with a uniform 1-cm three-dimensional margin around the surgical clips. The CTV was limited to 3 mm from the skin surface and 3 mm from the lung-chest wall interface. A second uniform, three-dimensional 1-cm margin was added to the CTV to obtain the planning target volume (PTV). The PTV was allowed to extend 4 mm inside the ipsilateral lung and was limited to 3 mm from the skin. The ipsilateral and contralateral breast, ipsilateral and contralateral lung, heart, and spinal cord were contoured as organs at risk.

All the regions of interest were contoured according to the International Commission on Radiation Units and Measurements reports 50 and 62 recommendations. No respiratory control was used.

Concerning the experimental Arm (accelerated partial breast irradiation), a dose of 30 Gy in five fractions at 6 Gy/fraction was prescribed.

The following constraints were adopted for plan optimization: PTV coverage: 100% of PTV covered by 95% of the prescribed dose (V28.5 = 100%); maximal dose to PTV <105% (31.5 Gy); minimal dose to PTV 28 Gy; uninvolved breast (i.e., ipsilateral breast without PTV): not >50% covered by a dose of >50% of the prescribed dose (V15 <50%); ipsilateral lung: not >20% covered by a dose >10 Gy (V10<20%); contralateral lung: not >10% covered by a dose >5 Gy (V5<10%); contralateral breast: maximal dose <1 Gy; heart: not >10% covered by a dose >3 Gy (V3 <10%).

ELIGIBILITY:
Inclusion Criteria:

* Age at presentation >40 y
* Tumor size <25 mm
* Wide excision or quadrantectomy with clear margins (>5 mm)
* Clips placed in tumor bed
* Full informed consent from patient

Exclusion Criteria:

* Cardiac dysfunction
* Forced expiratory volume in 1 second (FEV1) <1 L/m
* Extensive intraductal carcinoma
* Multifocal cancer
* Psychiatric problems
* Recurrent breast cancer

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2005-03; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Livi, Full Prof, Principal Investigator — Florence University; Icro Meattini, M.D., Principal Investigator — Azienda Ospedaliero-Universitaria Careggi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Livi L, Buonamici FB, Simontacchi G, Scotti V, Fambrini M, Compagnucci A, Paiar F, Scoccianti S, Pallotta S, Detti B, Agresti B, Talamonti C, Mangoni M, Bianchi S, Cataliotti L, Marrazzo L, Bucciolini M, Biti G. Accelerated partial breast irradiation with IMRT: new technical approach and interim analysis of acute toxicity in a phase III randomized clinical trial. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):509-15. doi: 10.1016/j.ijrobp.2009.04.070. Epub 2009 Aug 21. PMID 19700248
- [Result] Livi L, Meattini I, Marrazzo L, Simontacchi G, Pallotta S, Saieva C, Paiar F, Scotti V, De Luca Cardillo C, Bastiani P, Orzalesi L, Casella D, Sanchez L, Nori J, Fambrini M, Bianchi S. Accelerated partial breast irradiation using intensity-modulated radiotherapy versus whole breast irradiation: 5-year survival analysis of a phase 3 randomised controlled trial. Eur J Cancer. 2015 Mar;51(4):451-463. doi: 10.1016/j.ejca.2014.12.013. Epub 2015 Jan 17. PMID 25605582
- [Result] Meattini I, Saieva C, Marrazzo L, Di Brina L, Pallotta S, Mangoni M, Meacci F, Bendinelli B, Francolini G, Desideri I, De Luca Cardillo C, Scotti V, Furfaro IF, Rossi F, Greto D, Bonomo P, Casella D, Bernini M, Sanchez L, Orzalesi L, Simoncini R, Nori J, Bianchi S, Livi L. Accelerated partial breast irradiation using intensity-modulated radiotherapy technique compared to whole breast irradiation for patients aged 70 years or older: subgroup analysis from a randomized phase 3 trial. Breast Cancer Res Treat. 2015 Oct;153(3):539-47. doi: 10.1007/s10549-015-3565-2. Epub 2015 Sep 9. PMID 26350524
- [Derived] Meattini I, Marrazzo L, Saieva C, Desideri I, Scotti V, Simontacchi G, Bonomo P, Greto D, Mangoni M, Scoccianti S, Lucidi S, Paoletti L, Fambrini M, Bernini M, Sanchez L, Orzalesi L, Nori J, Bianchi S, Pallotta S, Livi L. Accelerated Partial-Breast Irradiation Compared With Whole-Breast Irradiation for Early Breast Cancer: Long-Term Results of the Randomized Phase III APBI-IMRT-Florence Trial. J Clin Oncol. 2020 Dec 10;38(35):4175-4183. doi: 10.1200/JCO.20.00650. Epub 2020 Aug 24. PMID 32840419
- [Derived] Becherini C, Meattini I, Livi L, Garlatti P, Desideri I, Scotti V, Orzalesi L, Sanchez LJ, Bernini M, Casella D, Nesi S, Nori J, Bianchi S, Pallotta S, Marrazzo L. External accelerated partial breast irradiation for ductal carcinoma in situ: long-term follow-up from a phase 3 randomized trial. Tumori. 2019 Jun;105(3):205-209. doi: 10.1177/0300891618811278. Epub 2018 Nov 26. PMID 30474504
- [Derived] Meattini I, Saieva C, Miccinesi G, Desideri I, Francolini G, Scotti V, Marrazzo L, Pallotta S, Meacci F, Muntoni C, Bendinelli B, Sanchez LJ, Bernini M, Orzalesi L, Nori J, Bianchi S, Livi L. Accelerated partial breast irradiation using intensity modulated radiotherapy versus whole breast irradiation: Health-related quality of life final analysis from the Florence phase 3 trial. Eur J Cancer. 2017 May;76:17-26. doi: 10.1016/j.ejca.2017.01.023. Epub 2017 Mar 3. PMID 28262584

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole Breast Irradiation (WBI) | Partial Breast Irradiation (APBI)
Started | 260 | 260
Completed | 260 | 246
Not Completed | 0 | 14
Not completed — Withdrawal by Subject | 0 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Breast Irradiation (WBI) | Partial Breast Irradiation (APBI) | Total
Number analyzed (Participants) | 260 | 260 | 520
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 158 | 142 | 300
  >=65 years | 102 | 118 | 220
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260 | 260 | 520
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 260 | 260 | 520

OUTCOME MEASURES:

1. Primary Outcome: Ipsilateral Breast Tumor Recurrence
Description: We defined local relapse (true recurrence) as the reappearance of the breast cancer in the index quadrant and ipsilateral breast tumours as any new breast cancer diagnosed in other quadrants of the same breast. The sum of local relapses and new ipsilateral breast tumours was defined as the ipsilateral breast tumour recurrence (IBTR). Locoregional tumour recurrence also included any recurrence in the ipsilateral axillary, supraclavicular, or internal mammary chain nodal regions.here we report the percentage of participants in each arm who experienced "Ipsilateral Breast Tumor Recurrence"
Time Frame: 5-year
Measure: Number; unit: percentage of participants
Arm/Group | Whole Breast Irradiation (WBI) | Partial Breast Irradiation (APBI)
Number analyzed (Participants) | 260 | 260
percentage of participants | 1.4 | 1.5

2. Secondary Outcome: Acute Skin Toxicity
Description: Acute skin toxicity ≥ grade 2, here we report the percentage of participants in each arm who experienced "Acute skin toxicity ≥ grade 2
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Whole Breast Irradiation (WBI) | Partial Breast Irradiation (APBI)
Number analyzed (Participants) | 260 | 260
percentage of participants | 37.7 | 2

3. Secondary Outcome: Excellent Cosmesis
Description: Physician-rated cosmesis, Cosmetic outcome was scored on the four-category Harvard Breast Cosmesis Scale. An excellent cosmetic result score was assigned when the treated breast looked like the contralateral one; a good cosmetic score was assigned for minimal but identifiable radiation effects of the treated breast; a fair score was used if significant radiation effects were readily observable; a poor score was used for severe sequelae due to radiation effects
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Whole Breast Irradiation (WBI) | Partial Breast Irradiation (APBI)
Number analyzed (Participants) | 260 | 260
percentage of participants | 89.6 | 95.1

ADVERSE EVENTS:
Time Frame: 5-years
Description: Acute and late skin toxicity, any grade
Arm/Group | Whole Breast Irradiation (WBI) | Partial Breast Irradiation (APBI)
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/246
Other Adverse Events (participants affected / at risk) | 173/260 | 49/246
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Whole Breast Irradiation (WBI) (N=260) | Partial Breast Irradiation (APBI) (N=246)
acute skin toxicity, any grade (Skin and subcutaneous tissue disorders) | 173 | 49 — Here we report total rate of acute skin toxicity in each arm of the study
late skin toxicity, any grade (Skin and subcutaneous tissue disorders) | 29 | 11 — Here we report rate of late skin toxicity in each arm of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No